CLINICAL TRIAL: NCT05701098
Title: Pivotal Study of the SonoMotion Break Wave™ (Trade Mark) System for the Comminution of Urinary Tract Stones
Brief Title: SOUND Pivotal Trial - (Sonomotion stOne comminUtion resoNance ultrasounD)
Acronym: SOUND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SonoMotion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0002
Record Dates: First submitted 2023-01-11; First posted 2023-01-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Kidney Stone; Urolithiasis; Nephrolithiasis; Renal Calculi; Kidney Calculi; Nephrolith; Urinary Calculi
Keywords: Kidney Stone; Urolithiasis; Nephrolithiasis; Renal Calculi; Kidney Calculi; Nephrolith; Urinary Calculi; Ultrasound therapy; Non-invasive; Extracorporeal
MeSH Terms: conditions — Kidney Calculi; Urolithiasis; Nephrolithiasis; Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Break Wave™ Procedure (Experimental): The subject will undergo the Break Wave procedure.
  Interventions: Device: Break Wave extracorporeal lithotripsy

INTERVENTIONS:
Device: Break Wave extracorporeal lithotripsy — The Break Wave device will be used to exert a low amplitude burst of ultrasound waves focused at the kidney stone. The primary components of the device include an ultrasound imaging system and a therapy probe driven by a high voltage generator. The probe will be placed on the patient's skin, the stone located via diagnostic ultrasound and up to 30 minutes of therapy will be delivered to the stone. The therapy probe accommodates coaxial alignment of an ultrasound imaging probe for treatment guidance.

SUMMARY:
The goal of this clinical trial is to test the Break Wave™ system in patients with upper urinary tract stones. The main question it aims to answer is whether the device is safe and effective in fragmenting (breaking) stones.

Participants will a) undergo the Break Wave™ procedure, b) have a telehealth visit at 2 weeks, and c) return for an imaging study at approximately 10 weeks post-procedure.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, single-arm (non-randomized) study to demonstrate the safety and effectiveness of breaking stones in the upper urinary tract using the SonoMotion Break Wave™ technology. Up to 116 patients will be screened to participate. Depending on the institution, the procedure may be performed in an outpatient hospital surgical environment, or in a non-surgical environment such as a clinic or office procedure room. Subjects will have a target stone diagnosed to be >4millimeter (mm) to 10 mm in size.

Safety will be measured by the adverse event occurrence, unplanned emergency department or clinic visits, and the need for further intervention. Effectiveness will be determined by the size of fragments identified at the 10 week follow-up imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects presenting with at least one stone apparent on radiographic imaging.
2. Target stone must be within the upper urinary tract.
3. Target stone is indicated for shock wave lithotripsy (SWL) treatment per American Urological Association (AUA) 2016 guidelines.
4. Target stone size is > 4 mm and ≤ 10 mm.
5. Subject is willing and able to provide informed consent and comply with the study protocol required follow up visits.
6. Target stone can be individually visualized from other stones.

Exclusion Criteria:

1. Subject has an acute untreated urinary tract infection or urosepsis.
2. Subject has an uncorrected bleeding disorder or coagulation abnormality.
3. Subject is confirmed to be or suspected to be pregnant.
4. Subject has a urinary tract obstruction distal to the stone.
5. Subject is receiving anticoagulants and is unable or not willing to cease the medication for the Break Wave procedure
6. Subject has stones that are not echogenically visible with ultrasound.
7. Subject belongs to a vulnerable group (prisoner, etc.).
8. Patients unwilling to comply with the follow-up protocol, including post-procedure radiographic imaging.
9. Subject is under 18 years of age.
10. Subject's anatomy limits ability to focus on or deliver Break Wave to the target stone (e.g. viable acoustic window).
11. Subject has a calcified abdominal aortic aneurysm or calcified renal artery aneurysms.
12. Subject has a solitary kidney.
13. Subject has a comorbidity risk(s) which, at the discretion of the physician, would make the subject a poor candidate for the Break Wave procedure, such as anatomical anomalies that may not be conducive to adequate stone fragment passage.
14. Subject is unable to read or comprehend the consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 10 +/- 2 weeks post final Break Wave procedure
  Proportion of subjects with a radiographic assessment of the target stone demonstrating either (i) stone free status (zero fragments) or (ii) the presence of only stone fragments small enough to pass spontaneously (≤ 4 mm).
Primary Safety Endpoint | During procedure and through 90 days post-procedure
  Occurrence of device and procedure related clinically significant or symptomatic hematoma (perirenal/intrarenal), urinary tract sepsis, or serious cardiac arrhythmia

SECONDARY OUTCOMES:
Secondary safety endpoint | During procedure and through 90 days post-procedure
  Occurrence of all device and procedure related adverse events (AEs), including serious adverse events (SAEs), and Unanticipated Adverse Device Effects (UADEs)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - University of California- San Diego, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - Kaiser Permanente, Santa Clara, California
  - Northwestern Medicine, Chicago, Illinois
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington, Seattle, Washington
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - St. Michael's Hospital, University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No